CLINICAL TRIAL: NCT05623215
Title: Comparing the Migration and Inducible Displacement Through RSA of the Cementless ATTUNE Rotating Platform and the Cementless LCS Rotating Platform Knee System; A Clinical Randomized Controlled RSA Follow-up Study
Brief Title: ALknee Follow-up Study of the Cementless ATTUNE Rotating Platform and the Cementless LCS Rotating Platform Knee System
Status: Active, not recruiting | Type: Observational
Sponsor: Spaarne Gasthuis (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Raymond Puijk, drs, Spaarne Gasthuis
Other Study IDs: NL82000.058.22
Record Dates: First submitted 2022-11-03; First posted 2022-11-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Total Knee Arthroplasty; Total Knee Replacement; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cementless ATTUNE: Cementless ATTUNE Rotating Platform Cruciate Sacrificing Knee System
  Interventions: Radiation: Radiographs of the knee for radiostereometric analysis (RSA)
- Cementless LCS: Cementless LCS rotating platform Cruciate Sacrificing Knee System
  Interventions: Radiation: Radiographs of the knee for radiostereometric analysis (RSA)

INTERVENTIONS:
Radiation: Radiographs of the knee for radiostereometric analysis (RSA) — RSA radiographs will be made 5 and 10 years after the total knee arthroplasty.

SUMMARY:
The cementless ATTUNETM Rotating Platform Knee system was compared in a single-blind, randomized RSA trial to its predecessor, the LCS rotating platform Knee System. In this previous study, 61 knees were subjected to RSA examinations at 1-day and 3, 6, 12 and 24 months postoperative. This study found a promising equal migration of both tibial components and a lesser migration of the femoral component of the ATTUNETM knee system after two years, although with a similar migration rate between year 1 and 2. this raises the question of whether the migration of the prostheses relative to each other will increase or remain the same in the long term. To examine this, a mid-and long-term RSA follow-up to measure migration is necessary. In addition, another new RSA measurement parameter has become known in recent years that may provide an indication of the bonding of the prosthesis to the bone at the time of measurement. This new parameter, called the Induced Displacement (ID) of a prosthesis, measures the position and orientation relative to the bone while the prosthesis is under different loading conditions (e.g., patient in supine or standing position). This means that a large measured difference between these different loading condition measurements would indicate that osseointegration of the prosthesis never occurred or is no longer present. To improve the understanding of the tendency of both prostheses to aseptic loosening after a mid- to long-term follow up, migration over time and inducible displacement analyses are necessary.

The primary objective of this study is to accurately compare mid- and long-term migration of two uncemented TKR prostheses. The secondary objectives of this study are to evaluate if inducible displacement can be used as a parameter to detect loose implants, and to compare inducible displacement, clinical and radiological outcome and patient-reported outcomes (PROMS) after a follow-up of 5 and 10 years of two uncemented TKR prostheses.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* The Patient participated in the initial study (NL58911.058.16) [1].
* The patient is capable of giving informed consent and expressing a willingness to comply with the study.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* The patient underwent a major revision TKR (exchange of the tibial or femoral component).
* The patient is unable or unwilling to sign the informed consent specific to this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In this study, all subjects that participated in the initial study (ALknee study - NL58911.058.16) will be asked to participate. All these patients underwent a TKA for symptomatic osteoarthritis of the knee in the period of August 2017 and March 2018 at the Department of Orthopaedics in the Spaarne Gasthuis, Hoofddorp, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline migration of the prostheses | 5 years post TKA
  Migration is measured and expressed in translations, rotations, and MTPM; MTPM is the point of the prosthesis that has moved most.
Ten year change from baseline migration of the prostheses | 10 years post TKA
  Migration is measured and expressed in translations, rotations and MTPM; MTPM is the point of the prosthesis that has moved most.

SECONDARY OUTCOMES:
Inducible displacement | 5 years post TKA
  The inducible displacement is defined as the difference in translation (MTPM) between a measurement without external force (e.g., supine position) and a measurement with external force (e.g., weight bearing) minus the measurement error.
Inducible displacement | 10 years post TKA
  The inducible displacement is defined as the difference in translation (MTPM) between a measurement without external force (e.g., supine position) and a measurement with external force (e.g., weight bearing) minus the measurement error.
EuroQol 5D-5L (EQ-5D-5L) | 5 year post TKA
  A patient reported outcome score for assessing mental well-being by using a score from 0 to 1, with 0 = worse and 1 = best.
EuroQol 5D-5L (EQ-5D-5L) | 10 year post TKA
  A patient reported outcome score for assessing mental well-being by using a score from 0 to 1, with 0 = worse and 1 = best.
Knee injury and Osteoarthritis Outcome Scale Physical Function Short-form (KOOS-PS) | 5 year post TKA
  A 7-item patient reported outcome score that measures daily physical functioning by using a score of 0 to 100, with 0 = no problems and 100 = extreme problems.
Knee injury and Osteoarthritis Outcome Scale Physical Function Short-form (KOOS-PS) | 10 year post TKA
  A 7-item patient reported outcome score that measures daily physical functioning by using a score of 0 to 100, with 0 = no problems and 100 = extreme problems.
Oxford-12 Knee Score (OKS) | 5 year post TKA
  A 12-item patient-reported outcome score to assess function and pain after total knee arthroplasty. The score uses a score of 0 to 48, with 0 = worse and 48 = best.
Oxford-12 Knee Score (OKS) | 10 year post TKA
  A 12-item patient-reported outcome score to assess function and pain after total knee arthroplasty. The score uses a score of 0 to 48, with 0 = worse and 48 = best.
Kujala Anterior Knee Pain Scale (AKPS) | 5 year post TKA
  A 13-item patient reported outcome score for assessing daily anterior knee pain, by using a score from 0 to 100, with 0 = having anterior knee pain with disabilities and 100 = no signs of anterior knee pain.
Kujala Anterior Knee Pain Scale (AKPS) | 10 year post TKA
  A 13-item patient reported outcome score for assessing daily anterior knee pain, by using a score from 0 to 100, with 0 = having anterior knee pain with disabilities and 100 = no signs of anterior knee pain.
Numeric Rating Scale (NRS) | 5 year post TKA
  A patient reported outcome score for assessing pain by using a likert scale from 0 to 10, with 0 = no pain and 10 = severe pain)
Numeric Rating Scale (NRS) | 10 year post TKA
  A patient reported outcome score for assessing pain by using a likert scale from 0 to 10, with 0 = no pain and 10 = severe pain)
Anchor questions | 5 year post TKA
  A patient reported outcome score for assessing change in functioning and pain since surgery.
  The outcome is evaluated by use of a likert scale from 1 to 7, with 1 = much deteriorated and 7 = much improved).
Anchor questions | 10 year post TKA
  A patient reported outcome score for assessing change in functioning and pain since surgery.
  The outcome is evaluated by use of a likert scale from 1 to 7, with 1 = much deteriorated and 7 = much improved).

OTHER OUTCOMES:
Complications | 5 year post TKA
  Complications during follow-up will be reported
Complications | 10 year post TKA
  Complications during follow-up will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Nolte, Prof. MD, Principal Investigator — Spaarne Gasthuis
Locations (1):
- Spaarne Gasthuis, Hoofddorp, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No